CLINICAL TRIAL: NCT00324662
Title: ADRIA - Belos A+ vs DR Clinical Investigation of Arrhythmia Discrimination
Brief Title: Study to Verify Proper Detection of Supraventricular Tachyarrhythmia With Single-Lead Dual-Chamber Implantable Cardioverter-Defibrillators (ADRIA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA044
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Tachyarrhythmia
Keywords: Implantable cardioverter-defibrillator; Ventricular tachyarrhythmia; Supraventricular tachyarrhythmia; Electric Countershock
MeSH Terms: conditions — Tachycardia; Tachycardia, Ventricular | interventions — Defibrillators, Implantable

INTERVENTIONS:
Device: Implantable cardioverter-defibrillator

SUMMARY:
A unique single-lead dual-chamber implantable cardioverter-defibrillator (ICD) system (produced by Biotronik, Germany) features a conventional electrode in the ventricle (anchored in the ventricular apex) and a floating electrode (ring on the lead body) in the atrium, capable of sensing atrial electrical signals. The purpose of this study is to determine whether this system detects a supraventricular tachyarrhythmia (e.g. atrial fibrillation, atrial tachycardia) in the equivalent manner as conventional dual-lead dual-chamber ICDs using two separate electrodes anchored in the ventricle and in the atrium, respectively.

DETAILED DESCRIPTION:
Supraventricular tachyarrhythmia (SVT) is the main cause of inappropriate therapy in patients with single-chamber implantable cardioverter-defibrillators (ICDs). To minimize inappropriate shock delivery, ICDs should sense both atrial and ventricular intracardiac signals. Dual-chamber ICDs are used for this purpose, but are associated with increased postoperative complications due to the implantation of a separate atrial lead. It has to be shown that a novel single-lead dual-chamber ICD-system with enhanced SVT discrimination can achieve the same specificity in discriminating SVT episodes as conventional dual-chamber ICD, without the disadvantage of the implantation of several leads. In this study patients eligible for dual-chamber ICD therapy who do not need atrial pacing will receive either a single-lead dual-chamber ICD (Belos A+ and Kainox A+ electrode) or a dual-lead dual-chamber ICD (Belos DR). SMART detection algorithm will be used in both study groups for discrimination between atrial and ventricular tachyarrhythmias. Atrial tachyarrhythmia episodes are facultatively induced in both groups at implantation or predischarge via a bipolar stimulation catheter. Induced episodes and the corresponding ICD intervention (detection and therapy or inhibition of therapy) are documented. Follow-ups are scheduled for 1, 3, 6 and 12 months after implantation. ICD intervention, particularly related to spontaneous SVT episodes, will be evaluated based on ICD diagnostic memory data interrogated at follow-up controls.

ELIGIBILITY:
Inclusion Criteria:

* ICD indication according to American College of Cardiology/American Heart Association (ACC/AHA) guidelines.
* Informed consent

Exclusion Criteria:

* Permanent atrial fibrillation
* Requirement for atrial pacing
* Patient is underage
* No signed patient agreement
* Patient life expectancy under 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Rate of correctly discriminated supraventricular tachyarrhythmia episodes (specificity)

SECONDARY OUTCOMES:
Complication rate (e.g. lead dislocation, lead fracture)
Duration of implantation
Electrode performance (P-/R-wave amplitudes, ventricular pacing threshold and impedance)
Sensitivity (rate of correctly discriminated episodes of ventricular fibrillation or ventricular tachycardia)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Niehaus, Prof. Dr. Med., Principal Investigator — Medizinische Hochschule Hannover, Abt. Kardiologie, Carl-Neuberg-Str. 1, 30625 Hannover, Germany
Locations (10):
- Germany (9):
  - Sana Klinikum Lichtenberg, Berlin
  - Charité-Universitätsmedizin Campus Benjamin Franklin, Med. Klinik II / Kardiologie, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH (Humboldt), Berlin
  - Kardiologische Praxis, Bonn
  - St. Johannes Hospital, Medizinische Klinik I, Dortmund
  - Georg-August-Universität, Universitätsklinikum Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Westfälische Wilhelms-Universität, Münster
  - Klinikum der Stadt Villingen Schwenningen GmbH, Villingen
- Kantonspital Basel, Abteilung für Kardiologie, Basel, Switzerland

REFERENCES:
- [Derived] Sticherling C, Zabel M, Spencker S, Meyerfeldt U, Eckardt L, Behrens S, Niehaus M; ADRIA Investigators. Comparison of a novel, single-lead atrial sensing system with a dual-chamber implantable cardioverter-defibrillator system in patients without antibradycardia pacing indications: results of a randomized study. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):56-63. doi: 10.1161/CIRCEP.110.958397. Epub 2010 Dec 14. PMID 21156772